CLINICAL TRIAL: NCT03448263
Title: Reduction of Post-endodontic Pain After Single-visit RCT Using Balanced Force and Two Reciprocating System When Intracanal Cryotherapy is Used.
Brief Title: Reduction of Post-endodontic Pain After RCT When Intracanal Cryotherapy is Used.
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, JORGE PAREDES VIEYRA D.D.S., MsC, PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Endo Pain 2018
Record Dates: First submitted 2018-02-15; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Post Operative Pain
Keywords: pain; post endodontic pain; root canal treatment
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Random Selection of instrumentation groups. Of the sample of 216 teeth, 72 were randomly assigned to the one of the 3 instrumentation methods. Treatment was performed by 3 experienced endodontists; each prepared 72 teeth, 24 per technique.
Who Masked: Participant, Investigator
Masking Description: Certified endodontists trained in the procedures, devices, and systems investigated took part in the research. All experts tracked a pre-established procedure for the Balanced Force technique, WaveOne, and Reciproc instrument systems.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group BF (Experimental): The root canals were cleaned and shaped using a #40 instrument for thin or curved canals and a #55 file for widespread canals.
  Interventions: Procedure: Balanced Force technique; Procedure: WaveOne technique; Procedure: Reciproc technique
- Group WON (Experimental): WaveOne files was used to prepare narrow, straight and curved canals, and a file (40.08) was used for large and wide canals.
  Interventions: Procedure: Balanced Force technique; Procedure: WaveOne technique; Procedure: Reciproc technique
- Reciproc instruments (Experimental): Reciproc instrument was used in thin and curved RC, and R40 files (40.06) were used in wide canals.
  Interventions: Procedure: Balanced Force technique; Procedure: WaveOne technique; Procedure: Reciproc technique

INTERVENTIONS:
Procedure: Balanced Force technique — Flex-R files sizes 15-45 taper .02 were used according to the technique on each tooth
Procedure: WaveOne technique — WaveOne instrument was used to prepare narrow, straight and curved canals, and file (40.08) was used for large canals.
  Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.
Procedure: Reciproc technique — Reciproc files were used in wide canals. Three in-and-out motions were used with lengths not beyond 3 mm in the three thirds of the canal until reaching the estimated WL.

SUMMARY:
The goal of this research was to relate the occurrence of post-endodontic pain after single-visit RCT using Balanced Force technique and two reciprocating system when cryotherapy is used. Methodology: All 216 patients had upper or lower molar, premolar or anterior teeth selected for conventional RCT for prosthetic reasons detected with only vital pulps. Of the sample of 216 teeth, were selected to the 3 instrumentation methods. For hand instrumentation, Balanced Force were used. All canals were clean and shaped with hand Flex-R files (fMoyco/Union Broach, York PA, USA). For mechanical shaping, all instruments were used with a micro motor (VDW, Munich Germany). WaveOne and Reciproc instruments. Final irrigation with cold (6oC) 17% EDTA served as a lubricant.

DETAILED DESCRIPTION:
Patient selection Two hundred and sixteen of 245 patients (119 women and 97 men) aged 18-65 years were incorporated in this research while 29 were excluded as not meeting the inclusion criteria. (Fig. 1). Sample size estimate was achieved according with a method for this specific purpose (Cochran's method, 1986). Therefore, the 56 teeth allocated to each group were adequate to confirm an essential sample size.

For hand instrumentation, the Balanced Force technique was used. All root canals were shaped with hand Flex-R files (Moyco/Union Broach, York PA, USA). Gates-Glidden drills (Dentsply Maillefer) sizes #2 and #3 were used at the orifice of the root canals. For mechanical preparations, all instruments were used with a micro motor (VDW Silver Motor, VDW, Munich Germany). Torque and rotation were preset for each Reciproc or WaveOne instrument. Rotary Ni-Ti instruments were used in continuous brushing rotary motion and reciprocating mode respectively.

Dentinal debris was eliminated from the file with a gauze, instantaneously to the instrument change (WaveOne) or after 2-3 in-and-out (pecking) movements (Reciproc) following the manufacturers' recommendations. Each root canal was irrigated with 2.5mL 2.6% NaOCl. Irrigation was performed using a 24-gauge needle (Max-I-Probe; Tulsa Dental, York, PA) and a 31-G NaviTip needle (Ultradent Products Inc, South Jordan, UT) when reaching the WL after each instrument insertion.

Group BF. For the Balanced Force group, the root canals were shaped and shaped using a #40 instrument for thin or curved canals and a #55 file for wide canals.

Group WON. For the WaveOne group, a file size 25/.08 was used to prepare narrow, straight and curved canals, and a file size 40/.08 was used for large and wide canals.

Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length.

Group REC. The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out pecking motions were used with an amplitude of not more than 3 mm until reaching the estimated working length.

ELIGIBILITY:
Inclusion Criteria:

The principal inclusion parameters were:

* absence of radiographic sign of apical periodontitis and a diagnosis of irreversible pulpitis (IP) established by affirmative response to hot and cold examinations.
* Thermal pulp examination was achieved by the corresponding author, and radiographic analysis was established by 3 certified endodontists.
* Clinical requirements were established on the next conditions: 1) The purposes and necessities of the research were spontaneously accepted. 2) Clinical Management was pointed to patients in physical and mental well-being. 3) All teeth had vital pulps and absence of apical periodontitis. 4) Positive thermal stimulation with EndoIce (Hygenic Corp, Akron, OH). 5) Teeth with enough coronal structure for rubber dam isolation. 6) No RCT done before the research. 7) No painkillers or antibiotics used 7 days' prior the clinical events started

Exclusion Criteria:

Exclusion parameters were:

* the necessity for retreatment
* gravidity
* impossibility to obtain patient's approval
* patients who didn't complete inclusion necessities
* a history of medication for chronic pain or those compromising the immune response
* patients younger than 18 years and the existence of mishaps or difficulties during RCT (calcified canals, impracticality of achieving AP in any canal).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the post-endodontic pain after single-visit After the root canal treatment with Balanced Force technique and two reciprocating system. | 24 hrs
  Post-endodontic pain was evaluated when the RCT developed with hand and rotary instruments

SECONDARY OUTCOMES:
Use of intracanal cryotherapy on post-endodontic pain after single-visit RC | 24 hrs
  A final irrigation after root canal treatment was made with cold 3cc of (6oC) 17% EDTA gently delivered to the WL using a cold (6oC) sterile metallic micro cannula.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Clemente Orozco, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729